CLINICAL TRIAL: NCT04507802
Title: Comparison of The Clinical Outcomes of Non-Invasive Ventilation by Helmet vs Facemask in Patients With Acute Respiratory Distress Syndrome
Brief Title: Helmet vs Face Mask in Patients With Acute Respiratory Distress Syndrome
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hamad Medical Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MRC-01-20-616
Record Dates: First submitted 2020-07-22; First posted 2020-08-11 (Actual); Last update posted 2020-08-11 (Actual); Status verified 2020-07

CONDITIONS: Acute Respiratory Distress Syndrome; Noninvasive Ventilation; Corona Virus Disease; Acute Respiratory Failure
MeSH Terms: conditions — Respiratory Distress Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Non invasive ventilation via helmet (Experimental): Patients who require noninvasive ventilation via Face mask for more than 8 hours will continue using noninvasive ventilation via facemask.
  Interventions: Device: Non invasive ventilation via helmet
- Non invasive ventilation via facemask (No Intervention): Patients assigned to the conventional ventilation group will continue noninvasive ventilation via facemask

INTERVENTIONS:
Device: Non invasive ventilation via helmet — Patients requiring long hours of noninvasive ventilation via facemask will switch to non-invasive ventilation using a helmet
  Arms: Non invasive ventilation via helmet

SUMMARY:
The objective of this study is to evaluate the efficacy of noninvasive ventilation with helmet in reducing endotracheal intubation rates in comparison with Noninvasive Ventilation (NIV) facemask among patients with Acute Respiratory Distress Syndrome (ARDS)

ELIGIBILITY:
Inclusion Criteria:

* Patients with (Acute Respiratory Distress Syndrome) ARDS as per Berlin definition
* Age: 18 and more

Exclusion Criteria:

* Patients with altered sensorium [Glasgow Coma Scale (GCS) less than 13]
* Pregnancy
* Hemodynamic instability
* Morbidly obese
* Patients with tracheostomy
* Severe acidosis [PH less than 7.15]
* Patients with glaucoma
* Patients with history of vertigo

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-08 (Estimated); Primary Completion 2021-05 (Estimated); Study Completion 2021-08 (Estimated)

PRIMARY OUTCOMES:
Need for Endotracheal Intubation | 6 weeks
  Number of patients requiring endotracheal intubation after application of helmet device

SECONDARY OUTCOMES:
Improvement in Oxygen Saturation | 2 weeks
  Improvement of oxygenation-defined as PaO2/FiO2 ≥ 200 or increase from baseline by 100
Ventilator-free Days | 28 days
  Duration of mechanical ventilation via endotracheal tube
Intensive Care Unit Length of Stay | 4 weeks
  Number of days admitted to intensive care unit
Overall Mortality | 90 days
  Death from any cause during hospitalization at time of enrollment
Need for Proning | up to 24 weeks
  Need for proning during the hospital stay
Intensive Care Unit Mortality | 28 days
  Death from any cause during ICU hospitalization at time of enrollment
Patient Tolerability | 28 days from randomization
  the degree to which overt adverse effects of a drug can be tolerated by a patient including feeding tolerance

CONTACTS AND LOCATIONS:
Overall Officials: Mohamad Y Khatib, MD, Principal Investigator — Hamad Medical Corporation
Locations (1):
- Hazm Mebaireek General Hospital (HMGH), Doha, Qatar

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Frutos-Vivar F, Nin N, Esteban A. Epidemiology of acute lung injury and acute respiratory distress syndrome. Curr Opin Crit Care. 2004 Feb;10(1):1-6. doi: 10.1097/00075198-200402000-00001. PMID 15166842
- [Background] Estenssoro E, Dubin A, Laffaire E, Canales H, Saenz G, Moseinco M, Pozo M, Gomez A, Baredes N, Jannello G, Osatnik J. Incidence, clinical course, and outcome in 217 patients with acute respiratory distress syndrome. Crit Care Med. 2002 Nov;30(11):2450-6. doi: 10.1097/00003246-200211000-00008. PMID 12441753
- [Background] Bellani G, Laffey JG, Pham T, Fan E, Brochard L, Esteban A, Gattinoni L, van Haren F, Larsson A, McAuley DF, Ranieri M, Rubenfeld G, Thompson BT, Wrigge H, Slutsky AS, Pesenti A; LUNG SAFE Investigators; ESICM Trials Group. Epidemiology, Patterns of Care, and Mortality for Patients With Acute Respiratory Distress Syndrome in Intensive Care Units in 50 Countries. JAMA. 2016 Feb 23;315(8):788-800. doi: 10.1001/jama.2016.0291. PMID 26903337
- [Background] ARDS Definition Task Force; Ranieri VM, Rubenfeld GD, Thompson BT, Ferguson ND, Caldwell E, Fan E, Camporota L, Slutsky AS. Acute respiratory distress syndrome: the Berlin Definition. JAMA. 2012 Jun 20;307(23):2526-33. doi: 10.1001/jama.2012.5669. PMID 22797452
- [Background] Ferguson ND, Fan E, Camporota L, Antonelli M, Anzueto A, Beale R, Brochard L, Brower R, Esteban A, Gattinoni L, Rhodes A, Slutsky AS, Vincent JL, Rubenfeld GD, Thompson BT, Ranieri VM. The Berlin definition of ARDS: an expanded rationale, justification, and supplementary material. Intensive Care Med. 2012 Oct;38(10):1573-82. doi: 10.1007/s00134-012-2682-1. Epub 2012 Aug 25. PMID 22926653
- [Background] Greene R, Lind S, Jantsch H, Wilson R, Lynch K, Jones R, Carvalho A, Reid L, Waltman AC, Zapol W. Pulmonary vascular obstruction in severe ARDS: angiographic alterations after i.v. fibrinolytic therapy. AJR Am J Roentgenol. 1987 Mar;148(3):501-8. doi: 10.2214/ajr.148.3.501. PMID 3492876
- [Background] Hess DR. Noninvasive ventilation for acute respiratory failure. Respir Care. 2013 Jun;58(6):950-72. doi: 10.4187/respcare.02319. PMID 23709194
- [Background] Berg KM, Clardy P, Donnino MW. Noninvasive ventilation for acute respiratory failure: a review of the literature and current guidelines. Intern Emerg Med. 2012 Dec;7(6):539-45. doi: 10.1007/s11739-012-0856-z. Epub 2012 Sep 28. PMID 23054404
- [Background] Carrillo A, Gonzalez-Diaz G, Ferrer M, Martinez-Quintana ME, Lopez-Martinez A, Llamas N, Alcazar M, Torres A. Non-invasive ventilation in community-acquired pneumonia and severe acute respiratory failure. Intensive Care Med. 2012 Mar;38(3):458-66. doi: 10.1007/s00134-012-2475-6. Epub 2012 Feb 9. PMID 22318634
- [Background] Thille AW, Contou D, Fragnoli C, Cordoba-Izquierdo A, Boissier F, Brun-Buisson C. Non-invasive ventilation for acute hypoxemic respiratory failure: intubation rate and risk factors. Crit Care. 2013 Nov 11;17(6):R269. doi: 10.1186/cc13103. PMID 24215648
- [Background] Antonelli M, Conti G, Esquinas A, Montini L, Maggiore SM, Bello G, Rocco M, Maviglia R, Pennisi MA, Gonzalez-Diaz G, Meduri GU. A multiple-center survey on the use in clinical practice of noninvasive ventilation as a first-line intervention for acute respiratory distress syndrome. Crit Care Med. 2007 Jan;35(1):18-25. doi: 10.1097/01.CCM.0000251821.44259.F3. PMID 17133177
- [Background] Schwartz AR, Kacmarek RM, Hess DR. Factors affecting oxygen delivery with bi-level positive airway pressure. Respir Care. 2004 Mar;49(3):270-5. PMID 14982647
- [Background] Patel BK, Wolfe KS, Pohlman AS, Hall JB, Kress JP. Effect of Noninvasive Ventilation Delivered by Helmet vs Face Mask on the Rate of Endotracheal Intubation in Patients With Acute Respiratory Distress Syndrome: A Randomized Clinical Trial. JAMA. 2016 Jun 14;315(22):2435-41. doi: 10.1001/jama.2016.6338. PMID 27179847
- [Derived] Khatib MY, Peediyakkal MZ, Elshafei MS, Elzeer HS, Ananthegowda DC, Shahen MA, Abdaljawad WI, Shaik KS, Kannappilly N, Mohamed AS, Soliman AA, Nashwan AJ. Comparison of the clinical outcomes of non-invasive ventilation by helmet vs facemask in patients with acute respiratory distress syndrome. Medicine (Baltimore). 2021 Jan 29;100(4):e24443. doi: 10.1097/MD.0000000000024443. PMID 33530249